CLINICAL TRIAL: NCT05978882
Title: Feasibility Study of Sentinel Navigation Surgery in Early Gastric Cancer Using Fluorescence (SENORITA4 Trial)
Brief Title: Feasibility Study of Sentinel Navigation Surgery in Early Gastric Cancer Using Fluorescence (SENORITA4)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Ajou University School of Medicine (Other); Chonnam National University Hospital (Other); Dongnam Institute of Radiological & Medical Sciences (Other); Gyeongsang National University Hospital (Other); Gyeongsang National University Changwon Hospital (Other); Samsung Medical Center (Other); Severance Hospital (Other); Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Hong Man Yoon, MD, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2023-0145
Record Dates: First submitted 2023-07-20; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Early Gastric Cancer
Keywords: Early gastric cancer; Sentinel lymph node; Fluorescence; Stomach-preserving surgery; Quality of life
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic sentinel navigation surgery (Experimental): compare the detection rate of sentinel lymph nodes to that of previous study (SENORITA1 trial)
  Interventions: Procedure: Laparoscopic sentinel navigation surgery using fluorescence

INTERVENTIONS:
Procedure: Laparoscopic sentinel navigation surgery using fluorescence — If the frozen biopsy of sentinel lymph nodes are all negative using fluorescence, stomach-preserving surgery is performed

SUMMARY:
SENORITA 1 trial showed laparoscopic sentinel lymph node biopsy and stomach preserving surgery in early gastric cancer can increase the quality of life. (Ryu KW et al. JCO 2022) The radioactive isotope is difficult to use because of the hazard of radiation and shortage of materials. The aim of this study is to investigate whether laparoscopic sentinel lymph node biopsy and stomach-preserving surgery using only fluorescence is feasible.

DETAILED DESCRIPTION:
1. Injection of Indocyanine Green (ICG)

   * Endoscopic injection of 0.25mg/ml of ICG on 4 sites around gastric cancer
   * Identification of sentinel basin using fluorescence laparoscopy
   * Laparoscopic sentinel basin dissection and identification of sentinel node at the back table
2. Surgical considerations

   * Conventional gastrectomy is performed if positive sentinel nodes are diagnosed in the frozen section.
   * If micrometastasis or isolated tumor cells in sentinel basin lymph nodes were diagnosed in permanent pathology, re-operation of conventional gastrectomy is not performed.
   * However, re-operation of conventional gastrectomy should be performed in case of macrometastasis, deep and lateral margin positive, more than pT2 lesion in the permanent pathology.

ELIGIBILITY:
Inclusion Criteria:

* single lesion of adenocarcinoma in preoperative endoscopic biopsy clinical stage T1N0 in the preoperative evaluation of endoscopy and computed tomography
* tumor size: less than 3cm
* location: 2cm far from the pylorus or cardia
* aged 20 to 80
* ECOG 0 or 1
* patient who signed the agreement
* patient who is suspected to underwent laparoscopic or robotic gastrectomy

Exclusion Criteria:

* indication of endoscopic submucosal resection
* inoperable due to poor cardiac, and pulmonary function
* pregnant
* having allergic reaction, previous upper abdominal surgery except laparoscopic cholecystectomy, previous radiation therapy to upper abdomen
* diagnosed as malignancy within 5 years except carcinoma in situ of cervix cancer and thyroid cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2023-08-17 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection rate of Sentinel lymph nodes | 15 days after operation
  number of patients whose sentinel nodes are detected / enrolled number of patients *100

SECONDARY OUTCOMES:
3 year disease free survival | 3 year after surgery
  A total of enrollment period is suspected to be three years and patients will be followed up for five years.
3 year overall survival rate | 3 year after surgery
  A total of enrollment period is suspected to be three years and patients will be followed up for five years.
3 year disease specific death rate | 3 year after surgery
  A total of enrollment period is suspected to be three years and patients will be followed up for five years.
3 year recurrence free survival rate | 3 year after surgery
  A total of enrollment period is suspected to be three years and patients will be followed up for five years.
scores of global health status scale, functional scales, and symptom scales/items of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) C30 and STO22 | 5 years
  Survey for quality of life will be performed regularly for three years after surgery. Measurement tool is the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) C30 and STO22. In EORTC QLQ C30, there are 1 global health status scale, 5 functional scales, and 9 symptom scales/items. EORTC QLQ STO22 includes 5 symptom scales and 4 single items. Each scale and item ranges 0 to 100. Higher score of global health status and functinoal scales indicate better quality of life and lower score of symptom scales indicates better quality of life. There is no summed score in these questionnaires.
5 year disease free survival rate | 5 years
  A total of enrollment period is suspected to be three years and patients will be followed up for five years. Therefore, we can complete data collection at five year later from when the last enrolled patients underwent intervention
5 year overall survival rate | 5 years
  A total of enrollment period is suspected to be three years and patients will be followed up for five years. Therefore, we can complete data collection at five year later from when the last enrolled patients underwent intervention
5 year disease specific death rate | 5 years
  A total of enrollment period is suspected to be three years and patients will be followed up for five years. Therefore, we can complete data collection at five year later from when the last enrolled patients underwent intervention
5 year recurrence free survival rate | 5 years
  A total of enrollment period is suspected to be three years and patients will be followed up for five years. Therefore, we can complete data collection at five year later from when the last enrolled patients underwent intervention

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Dongnam Inst. of Radiological & Medical Science, Busan, Gijang-gun
  - Gyeongsang National University Hospital, Gyeongsang, Gingu-si
  - Sevrance Hospital, Seoul, Sinchon
  - Ajou University Medical Center, Gyeonggi-do, Suwon-si
  - Gyeongsang National University Changwon Hospital, Changwon
  - Samsung Medical Center, Seoul
  - Soon Chun Hyang University Hospital Bucheon, Seoul